CLINICAL TRIAL: NCT00043550
Title: Efficacy of Dynamic Therapy Versus Selective Serotonin Reuptake Inhibitor for Depression
Brief Title: Treatments for Depression: Drug Versus Psychotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH061410 (NIH); R01MH061410 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Sertraline/Venlafaxine (Experimental): Participants receive sertraline for the first 8 weeks. Participants will receive venlafaxine if they do not respond to sertraline by week 8
  Interventions: Drug: Sertraline; Drug: Venlafaxine
- 2 Supportive Expressive Therapy (Active Comparator): Participants will receive supportive-expressive psychotherapy.
  Interventions: Behavioral: Supportive Expressive Therapy
- 3 Pill Placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Drug: Pill Placebo

INTERVENTIONS:
Behavioral: Supportive Expressive Therapy — The aim of supportive-expressive psychotherapy is to help patients understand the causes of relationship conflicts in the context of a supportive relationship.
  Arms: 2 Supportive Expressive Therapy
Drug: Sertraline — Participants will receive sertraline.
  Other Names: Zoloft
  Arms: 1 Sertraline/Venlafaxine
Drug: Pill Placebo — Participants will receive a pill placebo.
  Arms: 3 Pill Placebo
Drug: Venlafaxine — Participants will receive venlafaxine.
  Other Names: Effexor
  Arms: 1 Sertraline/Venlafaxine

SUMMARY:
This 4-8 month study, with a 2-year follow up period, will compare sertraline (Zoloft®), venlafaxine (Effexor®), supportive-expressive psychotherapy, and placebo to determine which is more effective in treating major depression.

DETAILED DESCRIPTION:
MDD is one of the most prevalent psychiatric disorders. Different forms of psychotherapy for depression have been found effective. This study compares a form of dynamic psychotherapy called supportive-expressive psychotherapy to medication and to placebo.

Participants are evaluated on 2 occasions, 1 week apart, before they are randomly assigned to receive either supportive-expressive psychotherapy, sertraline (Zoloft) (followed by venlafaxine [Effexor] if patients do not respond to sertraline), or placebo. The active phase of treatment lasts 4 months. The frequency of patients' visits depends on the assigned treatment.

Patients who are randomized to receive medication or placebo are initially seen on a weekly basis, then less often, depending on the rate of symptomatic improvement. Patients who are randomized to psychotherapy are seen twice a week for the first 4 weeks, then once a week for the remaining 12 weeks. Outcome is monitored at week 2,4,6,7,8, 12, 15 and 16. At the end of the first 16 weeks of treatment, patients are thoroughly evaluated. Those who have responded to treatment are assigned to a continuation phase and are seen once a month for another 16 weeks. At the end of the 16-week continuation phase, patients are again evaluated and all treatments are stopped. Follow-up continues every 3 months for up to 2 years to ensure that the patients' depression remains under control.

ELIGIBILITY:
Inclusion criteria:

* Major Depressive Disorder diagnosis

Exclusion criteria:

* Psychotic or bipolar disorder diagnosis
* Substance dependence in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2001-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Barber, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Barber JP, Muenz LR. The role of avoidance and obsessiveness in matching patients to cognitive and interpersonal psychotherapy: empirical findings from the treatment for depression collaborative research program. J Consult Clin Psychol. 1996 Oct;64(5):951-8. doi: 10.1037//0022-006x.64.5.951. PMID 8916624
- [Derived] Kuprian N, Aafjes-van Doorn K, Gutterman D, Barber JP. Therapeutic immediacy in psychodynamic psychotherapy for depression: A mixed-method study. Psychotherapy (Chic). 2022 Dec;59(4):554-566. doi: 10.1037/pst0000452. Epub 2022 Aug 1. PMID 35913883
- [Derived] Solomonov N, Falkenstrom F, Gorman BS, McCarthy KS, Milrod B, Rudden MG, Chambless DL, Barber JP. Differential effects of alliance and techniques on Panic-Specific Reflective Function and misinterpretation of bodily sensations in two treatments for panic. Psychother Res. 2020 Jan;30(1):97-111. doi: 10.1080/10503307.2019.1585591. Epub 2019 Mar 1. PMID 30821630
- [Derived] Solomonov N, McCarthy KS, Gorman BS, Barber JP. The Multitheoretical List of Therapeutic Interventions - 30 items (MULTI-30). Psychother Res. 2019 Jul;29(5):565-580. doi: 10.1080/10503307.2017.1422216. Epub 2018 Jan 16. PMID 29336228
- [Derived] Zilcha-Mano S, Keefe JR, Chui H, Rubin A, Barrett MS, Barber JP. Reducing Dropout in Treatment for Depression: Translating Dropout Predictors Into Individualized Treatment Recommendations. J Clin Psychiatry. 2016 Dec;77(12):e1584-e1590. doi: 10.4088/JCP.15m10081. PMID 28086005
- [Derived] Zilcha-Mano S, Dinger U, McCarthy KS, Barrett MS, Barber JP. Changes in well-being and quality of life in a randomized trial comparing dynamic psychotherapy and pharmacotherapy for major depressive disorder. J Affect Disord. 2014 Jan;152-154:538-42. doi: 10.1016/j.jad.2013.10.015. Epub 2013 Oct 16. PMID 24176534
- [Derived] Barber JP, Barrett MS, Gallop R, Rynn MA, Rickels K. Short-term dynamic psychotherapy versus pharmacotherapy for major depressive disorder: a randomized, placebo-controlled trial. J Clin Psychiatry. 2012 Jan;73(1):66-73. doi: 10.4088/JCP.11m06831. Epub 2011 Nov 29. PMID 22152401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 374 individuals, ages 18 to 70 years, were recruited through advertisements on public transportation, free news publications, area physicians, and outpatient clinics during the period of 2001-2006.
Pre-assignment Details: Individuals not meeting MDD diagnostic criteria11 using the Structured Clinical Interviews for DSM-IV12 or scoring less than 14 on the 17-item Hamilton Rating Scale for Depression (HRSD)13,14 at two evaluations one week apart were excluded (n=88).
Groups:
- 1 Sertraline: Participants receive sertraline.
  Sertraline : Participants will receive sertraline.
- 2 Supportive-expressive Psychotherapy: Participants will receive supportive-expressive psychotherapy.
  Supportive Expressive Therapy : The aim of supportive-expressive psychotherapy is to help patients understand the causes of relationship conflicts in the context of a supportive relationship.
- 3 Pill Placebo: Participants receive placebo.
  Pill Placebo : Participants will receive a pill placebo.
Period: Overall Study
Arm/Group | 1 Sertraline | 2 Supportive-expressive Psychotherapy | 3 Pill Placebo
Started | 55 | 51 | 50
Week 8 Completed | 35 | 40 | 35
Completed | 33 | 39 | 30
Not Completed | 22 | 12 | 20
Not completed — Withdrawal by Subject | 22 | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Sertraline | 2 Supportive-expressive Psychotherapy | 3 Pill Placebo | Total
Number analyzed (Participants) | 55 | 51 | 50 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 51 | 50 | 156
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (12.5) | 36.2 (12.2) | 38.3 (12.0) | 37.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 31 | 92
  Male | 25 | 20 | 19 | 64
Region of Enrollment [Number; unit: participants]
  United States | 55 | 51 | 50 | 156

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression-17 Item
Description: Hamilton Rating Scale for Depression (HRSD) (Hamilton, 1960). We used the 17-item version of the 27-item HRSD, a measure of depression severity. The Structured Interview Guide was used to conduct the interviews (SIGH-D; Williams, 1988). The reliability and validity of the HRSD are well documented (Rabkin & Klein, 1987). Interjudge reliability as assessed by interclass correlations was .92 in our sample. Total 17-item scores could range from 17-48 with higher scores indicating greater distress.
Time Frame: symptoms assessed during past 7 days, measure taken at baseline, week 8 and week 16
Population: Numbers vary from consented due to dropout prior to start of study. 156 patients consented and randomized. 11 patients did not complete at least one post-randomization measure and were therefore not included in these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Sertraline | 2 Supportive-expressive Psychotherapy | 3 Pill Placebo
Number analyzed (Participants) | 51 | 46 | 48
units on a scale
  Initial HRSD-17 | 19.0 (3.4) | 19.9 (3.9) | 19.4 (3.7)
  Mid-treatment HRSD-17 | 13.9 (7.2) | 12.5 (6.9) | 12.7 (6.8)
  LOCF HRSD-17 | 14.2 (7.6) | 14.5 (8.3) | 14.3 (7.6)
Statistical Analysis 1: Comparison: 1 Sertraline vs 2 Supportive-expressive Psychotherapy vs 3 Pill Placebo; Comparison of conditions; Test type: Superiority — The proposed sample size had at least 80% power to detect effect sizes of 0.36 between the two active treatment conditions and placebo during the active phase. These power calculations were based on a priori values of within-subject correlation of 0.50, 10% attrition, and 6 assessment points; p = .95, HLM — Overall significant effect for treatment, as well as the two moderating effects, used a Bonferroni-corrected alpha level of 0.0167 (0.05/3); Slope = 1
Statistical Analysis 2: Comparison: 1 Sertraline vs 2 Supportive-expressive Psychotherapy vs 3 Pill Placebo; effects of conditions over time; Test type: Superiority; p < .0001, HLM
Statistical Analysis 3: Comparison: 1 Sertraline vs 3 Pill Placebo; Test type: Superiority; Slope = .03, 95% CI 2-sided [-.35 to .41]
Statistical Analysis 4: Comparison: 2 Supportive-expressive Psychotherapy vs 3 Pill Placebo; Test type: Superiority; Slope = .06, 95% CI 2-sided [-.33 to .45]

ADVERSE EVENTS:
Arm/Group | 1 Sertraline | 2 Supportive-expressive Psychotherapy | 3 Pill Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/55 | 1/51 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Sertraline (N=55) | 2 Supportive-expressive Psychotherapy (N=51) | 3 Pill Placebo (N=50)
passive suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — patient reported taking 4.5 mg of alprazolam . An hour later he took venlafaxine 187.5 mg, methylphenidate 30mg, and oxycodone 5mg with acetominophen. Patient was taken to the hospital ER and released without medical intervention.

LIMITATIONS AND CAVEATS:
Two limitations are the relatively high level of attrition and small sample size for specific combinations within our moderation analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No